CLINICAL TRIAL: NCT01021137
Title: Vestibular Consequences of Blast-related Mild Traumatic Brain Injury
Brief Title: Vestibular Consequences of Blast-related Mild Traumatic Brain Injury (TBI)
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C6841-R
Record Dates: First submitted 2009-11-24; First posted 2009-11-26 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Dizziness; Brain Injury
Keywords: vestibular function tests; postural balance; neuroimaging
MeSH Terms: conditions — Dizziness; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- TBI & Blast: OEF/OIF Veterans complaining of dizziness and/or imbalance with history of blast exposure and a diagnosis of mild TBI
- Blast Only: OEF/OIF Veterans complaining of dizziness and/or imbalance with history of blast exposure without TBI
- TBI Only: OEF/OIF Veterans complaining of dizziness and/or imbalance with a history of mild TBI and no blast exposure
- Healthy Controls: Age and gender matched control participants with no complaints of dizziness and/or imbalance or history of TBI or blast exposure
- Excluded: Participants who did not meet inclusion criteria, did not return to complete evaluation, and/or were excluded from data analysis.

SUMMARY:
The purpose of this project is to determine the effects of mild traumatic brain injury and blast exposure on the inner ear balance and central nervous systems.

DETAILED DESCRIPTION:
The goal of this project is to determine the effects of mild traumatic brain injury (mTBI) and blast exposure on the vestibular system and CNS. Dizziness and balance disorders are common symptoms associated with mTBI or head injury. Numerous studies have provided significant evidence that mTBI or head injury can cause damage to the vestibular system; however, most have limited the vestibular evaluation to assessment of horizontal semicircular canal function. Recently, methods have been developed to assess otolith function, and there is some evidence that head injury may affect the otolith organs to a greater degree than the semicircular canals.

mTBI has been called the signature condition of Veterans returning from Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF), and the cause is often related to blast exposure from improvised explosive devices, mortars or rocket-propelled grenades. Some investigators have presumed that dizziness and balance disorders following blast exposure are related to CNS damage caused by the TBI rather than the pressure wave from the blast injury. Thus, most research has focused on the vestibular consequences of TBI (or head injury), and there is limited data on the effects of blast exposure on vestibular function or balance. Recently, magnetic resonance imaging techniques have been developed that may allow for testing the assumption that the symptoms of dizziness or imbalance related to head injury or blast exposure are often due to central vestibular or CNS involvement.

Specific aims of this project are to determine the effect of mTBI and blast exposure on (1) peripheral vestibular system function (specifically, horizontal semicircular canal function, and otolith organ function), (2) central vestibular/CNS function, (3) postural stability, and (4) dizziness-related quality of life. Four subject groups will include Veterans complaining of dizziness/imbalance with (1) a history of blast exposure, (2) with mTBI, (3) with blast exposure and mTBI, and (4) a control group. Each subject will undergo tests of horizontal semicircular canal function (caloric and rotary chair), tests of otolith function (vestibular evoked myogenic potentials, subjective visual vertical), central vestibular function/CNS function (ocular motor tests, diffusion tensor and susceptibility weighting imaging), gait and balance testing, and the Dizziness Handicap Inventory.

ELIGIBILITY:
Inclusion Criteria:

* Complaint of dizziness and/or imbalance
* History of blast exposure
* Diagnosis of mild traumatic brain injury

Exclusion Criteria:

* Prior history of vestibular or neurological disorder
* Presence of internal metal
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: OEF/OIF Veterans
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faith Akin, PhD, Principal Investigator — Mountain Home VA Medical Center James H. Quillen VA Medical Center, Mountain Home, TN
Locations (1):
- Mountain Home VA Medical Center James H. Quillen VA Medical Center, Mountain Home, TN, Mountain Home, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 140 Veterans were recruited for this study. Participants included Operation Enduring Freedom/Operation Iraqi Freedom (OEF/OIF) Veterans and healthy, age & gender matched controls. Veteran participants had a history of traumatic brain injury (TBI), blast exposure, or both.
Pre-assignment Details: Six participants were consented to participate in the study, but did not return to complete the protocol. Case history was not collected and therefore, the participants could not be assigned to any of the study groups.
Groups:
- Healthy Controls: Age and gender matched control subjects with no complaints of dizziness and/or imbalance or history of TBI or blast exposure
Period: Overall Study
Arm/Group | TBI & Blast | Blast Only | TBI Only | Healthy Controls
Started | 62 | 20 | 11 | 41
Completed | 52 | 16 | 9 | 32
Not Completed | 10 | 4 | 2 | 9
Not completed — Lost to Follow-up | 9 | 4 | 2 | 6
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants differs from the number of participants assigned to the groups due to participants being lost to follow-up and being withdrawn from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | TBI & Blast | Blast Only | TBI Only | Healthy Controls | Total
Number analyzed (Participants) | 52 | 16 | 9 | 32 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 51 | 16 | 9 | 32 | 108
  >=65 years | 1 | 0 | 0 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (9.9) | 40.5 (10.5) | 39.7 (10.9) | 31.2 (9.8) | 35.9 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 4 | 7
  Male | 51 | 15 | 8 | 28 | 102
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 16 | 9 | 32 | 109

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Vestibular Function (Vestibulo-ocular Reflex/Semicircular Canal): Caloric Weakness
Description: The caloric weakness was determined using monothermal warm inter-ear difference (MWIED) which was calculated as: (|RW| - |LW| )/( |RW| + |LW|) x 100, where RW = the maximum slow phase velocity (SPV) of nystagmus induced by warm water irrigation in the right ear and LW = the maximum SPV of nystagmus induced by warm water irrigation in the left ear. For participants with MWIED > 10, then cool caloric irrigation was also performed and caloric weakness was determined using a bithermal inter-ear difference (BIED) calculated as: (|RW| + |RC|) - (|LW| + |LC|) / (|RW| + |RC| + |LW| + |LC|) x 100, where RC = maximum SPV of nystagmus induced by cool water irrigation in the right ear and LC = maximum SPV of nystagmus induced by cool water irrigation in the left ear.
Time Frame: up to 30 minutes
Population: Caloric weakness could not be obtained from 1 participant in the Blast Only group and 2 participants in the Healthy Control group.
Measure: Mean (Standard Deviation); unit: percentage of caloric weakness
Arm/Group | TBI & Blast | Blast Only | TBI Only | Healthy Controls
Number analyzed (Participants) | 52 | 15 | 9 | 30
percentage of caloric weakness | 8.8 (8.5) | 14.7 (20.8) | 12.3 (5.6) | 7.1 (6.0)

2. Primary Outcome: Rotary Chair Slow Harmonic Acceleration (SHA) Gain
Description: Rotary chair slow harmonic acceleration (SHA) vestibulo-ocular reflex (VOR) gain at 0.01 Hz was used as a measure of peripheral vestibular function (VOR/horizontal semicircular canal). VOR gain is defined as the ratio of the slow component velocity eye movement (output) to the velocity of the head movement (input).
Time Frame: up to 30 minutes
Population: Rotary chair slow harmonic acceleration (SHA) VOR gain at 0.01 Hz was not evaluated in 1 participant in the TBI & Blast group.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | TBI & Blast | Blast Only | TBI Only | Healthy Controls
Number analyzed (Participants) | 51 | 16 | 9 | 32
Unitless | .4 (.1) | .4 (.1) | .4 (.1) | .4 (.1)

3. Primary Outcome: Peripheral Vestibular Function (Saccular-collic Pathway): Cervical Vestibular Evoked Potential (cVEMP)
Description: Air-conducted cervical vestibular evoked potential (cVEMP) inter-ear amplitude asymmetry ratio was used as a measure of otolith organ function (saccular-collic pathway). Inter-ear amplitude asymmetry ratio was calculated as: [(|L_P1-N1| - |R_P1-N1|)/ (|L_P1-N1| + |R_P1-N1|)] x100, where L_P1-N1 = peak-to-peak cVEMP amplitude of the left side and R_P1-N1 = peak-to-peak cVEMP amplitude of the right side. The amplitudes were calculated from cVEMP responses at a stimulus intensity of 120 dB peakSPL. The criterion for abnormal cVEMP was defined as an absent cVEMP or a corrected cVEMP amplitude asymmetry ratio greater than or equal to 40%, either of which would indicate a unilateral vestibular loss. A bilateral vestibular loss was indicated by absent cVEMPs bilaterally.
Time Frame: Up to 30 minutes
Population: Cervical VEMP could not be evaluated on 2 participants in the TBI & Blast group and 3 participants in the Blast Only group.
Measure: Mean (Standard Deviation); unit: percentage of inter-ear asymmetry
Arm/Group | TBI & Blast | Blast Only | TBI Only | Healthy Controls
Number analyzed (Participants) | 49 | 13 | 9 | 32
percentage of inter-ear asymmetry | 26.1 (26.2) | 31.2 (32.3) | 45.1 (36.5) | 20.1 (15.9)

4. Primary Outcome: Rotary Chair Slow Harmonic Acceleration (SHA) Phase
Description: Rotary chair slow harmonic acceleration (SHA) vestibulo-ocular reflex (VOR) phase at 0.01 Hz was used as a measure of peripheral vestibular function (VOR/horizontal semicircular canal). The phase is the timing difference between the velocity of head movement and the slow-phase eye velocity. This parameter is normalized for a full cycle of a sinusoid (360 degrees) and presented in an angular unit of degrees rather than a unit of time. For perfectly compensatory eye movements the phase is 0 degrees, meaning there is no difference between the actual eye velocity and the ideal VOR (by convention, degrees is added to the phase so that the comparison is based on the ideal VOR responses instead of the actual head motion).
Time Frame: Up to 30 minutes (SHA phase is obtained simultaneously with SHA gain)
Population: Rotary chair slow harmonic acceleration (SHA) phase at 0.01 Hz was not calculated for 2 participants in the TBI & Blast group and 1 participant in the Blast Only group. Phase at 0.01 Hz could not be calculated for individuals with bilateral vestibular loss.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | TBI & Blast | Blast Only | TBI Only | Healthy Controls
Number analyzed (Participants) | 49 | 15 | 9 | 32
degrees | 41.3 (8.1) | 40.1 (6.4) | 40.1 (8.8) | 42.2 (8.3)

5. Primary Outcome: Peripheral Vestibular Function (Utricular-ocular Pathway): Ocular Vestibular Evoked Potential (oVEMP)
Description: Bone-conducted ocular vestibular evoked potential (oVEMP) inter-ear amplitude asymmetry ratio was used as a measure of otolith organ function (utricular-ocular pathway). Inter-ear amplitude asymmetry ratio was calculated as: [(|L_N1-P1| - |R_N1-P1|)/ (|L_N1-P1| + |R_N1-P1|)] x100, where L_N1-P1 = peak-to-peak oVEMP amplitude of the left eye/right ear and R_N1-P1 = peak-to-peak oVEMP amplitude of the right eye/left ear. The oVEMP is a contralateral response; therefore, recordings from the left eye reflect the response of the right ear and vice versa. The amplitudes were calculated from oVEMP responses at a stimulus intensity of 155 dB peakFL. The criterion for abnormal oVEMP was defined as an absent oVEMP or a corrected oVEMP amplitude asymmetry ratio greater than or equal to 40%, either of which would indicate a unilateral vestibular loss. A bilateral vestibular loss was indicated by absent oVEMPs bilaterally.
Time Frame: Up to 20 minutes
Population: Ocular VEMP could not be obtained from 4 participants from the TBI & Blast group.
Measure: Mean (Standard Deviation); unit: percentage of inter-aural asymmetry
Arm/Group | TBI & Blast | Blast Only | TBI Only | Healthy Controls
Number analyzed (Participants) | 48 | 16 | 9 | 32
percentage of inter-aural asymmetry | 22.0 (21.2) | 15.7 (14.3) | 39.1 (28.3) | 18.0 (14.6)

6. Secondary Outcome: Central Vestibular/Central Nervous System (CNS) Function: Visual Fixation Suppression
Description: Visual fixation suppression was used as a measure of central vestibular/CNS function. Visual fixation suppression is a measure of vestibulo-ocular reflex (VOR) gain obtained during visual fixation at 0.16 Hz slow harmonic acceleration on the rotary chair. VOR gain was defined as the ratio of the slow component velocity eye movement (output) to the velocity of the head movement (input). Visual fixation suppression was considered normal if VOR gain is suppressed > 50% with visual fixation compared to no fixation.
Time Frame: 1 minute
Population: VOR gain during a visual fixation task and 0.16 Hz could not be obtained on 2 participants in the TBI & Blast group and 3 participants in the Blast Only group.
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | TBI & Blast | Blast Only | TBI Only | Healthy Controls
Number analyzed (Participants) | 49 | 13 | 9 | 32
unitless | 0.069 (0.049) | 0.058 (0.034) | 0.059 (0.034) | 0.065 (0.041)

7. Secondary Outcome: Postural Stability: Sensory Organization Test (SOT)
Description: This measure is the composite equilibrium score from six conditions of the sensory organization test obtained with the Neurocom Equitest. Results of the SOT were calculated based on maximum peak-to-peak anterior-posterior sway expressed as an equilibrium score ranging from 0 to 100, with 0 indicating loss of balance (i.e., required support of harness, took a step, touched walls for support or opened eyes in eyes closed conditions) and 100 indicating perfect stability. The outcome measure was the equilibrium composite score and was calculated by the software as the weighted average of the equilibrium scores for the six conditions. For ages 18-59 years, the normative value (mean - 1.67 SD) for the composite score is at least 70 (NeuroCom, 2011).
Time Frame: Up to 20 minutes
Population: The composite equilibrium score of the sensory organization test was not obtained for 4 participants in the TBI & Blast group, 2 participants in the Blast Only group and 2 participants in the Healthy Control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TBI & Blast | Blast Only | TBI Only | Healthy Controls
Number analyzed (Participants) | 48 | 14 | 9 | 30
units on a scale | 65 (18.8) | 62 (19.3) | 61 (16.1) | 81 (5.1)

8. Secondary Outcome: Dizziness Handicap Inventory
Description: The Dizziness Handicap Inventory (DHI) was used as a quality of life measure.The DHI measures the subject's self-perceived dizziness. The scale has 25 questions with 3 possible answers each: "Yes" = 4 points, "Sometimes" = 2 points, and "No" = 0 points. The minimum number of points that a subject can score is 0 and the maximum number of points is 100. The subject's self-perceived dizziness is reported as a percentage with a range of 0-100%, and is calculated by: subject's total number of points/maximum number of points (100) x 100%. The higher the score on the DHI, the worse a patient's self-perceived dizziness.
Time Frame: Up to 10 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TBI & Blast | Blast Only | TBI Only | Healthy Controls
Number analyzed (Participants) | 52 | 16 | 9 | 32
score on a scale | 48.7 (23.1) | 48.6 (25.5) | 41.6 (15.7) | 0 (0)

ADVERSE EVENTS:
Arm/Group | TBI & Blast | Blast Only | TBI Only | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/20 | 0/11 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/20 | 0/11 | 0/41
Other Adverse Events (participants affected / at risk) | 0/62 | 0/20 | 0/11 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes